CLINICAL TRIAL: NCT01091311
Title: Phase IV Multicentric Study, 30 Patients Suffering of Meibomian Glands Dysfunction.
Brief Title: Evaluation of Satisfaction Regarding Patient's Management of Ocular Surface Diseases
Acronym: ESPOIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT2420-PIV-CE-01/10; N° RCB 2010-A00017-32 (Other: AFSSAPS)
Record Dates: First submitted 2010-03-19; First posted 2010-03-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Eyelid Diseases
Keywords: Meibomian Gland Dysfunction
MeSH Terms: conditions — Eyelid Diseases; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Blephasteam — Eye lid warming goggles

SUMMARY:
Multicentric study, open label, uncontrolled phase IV in 30 patients with meibomian glands dysfunction .

Its objective is to Collect information from patients and ophthalmologists specialized in ocular surface and eyelids to anticipate how Blephasteam ® can be optimized.

This study involves 2 visits, visit of Inclusion, J0, then end of study visit, D21.

Between the two visits patients will be treated with Blephasteam ® for 21 days (up to two uses per day) and complete a questionnaire every two days during the first week and then once a week the next two weeks.

ELIGIBILITY:
* Signed and dated informed consent.
* Male or female up to 4 years old.
* Known and treated symptomatic Meibomian Gland Diseases, and/or Dry Eye related to MGDs stable since at least a month.
* Without any active pathology requiring a change in ocular treatments within the last month before inclusion.
* Best corrected far visual acuity (VA) > 1/10

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Baudouin, Professor, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts; Frédéric Chiambaretta, Professor, Principal Investigator — University Hospital, Clermont-Ferrand; Serge Doan, Doctor, Principal Investigator — Hopital Bichat
Locations (3):
- France (3):
  - HÃ´pital Gabriel Montpied, Clermont-Ferrand
  - C.H.N.O des XV-XX, Paris
  - Hôpital Bichat - Claude Bernard, Paris